CLINICAL TRIAL: NCT05773521
Title: Comparative Retrospective Study on the Different Analgesic Modalities Used for Single-incision Laparoscopic Appendectomy
Brief Title: Peri-operative Analgesia for Single-incision Laparoscopic Appendectomy
Acronym: PAMAL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-124
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Appendicitis
Keywords: appendectomy; single-site laparoscopy; analgesia; pain; peri-operative management
MeSH Terms: conditions — Appendicitis; Agnosia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SILAP patients: This cohort is composed by all pediatric patients operated on for SILAP between January 1st, 2012 and August 31, 2022.
  Interventions: Procedure: SILAP (single incision laparoscopic appendectomy)

INTERVENTIONS:
Procedure: SILAP (single incision laparoscopic appendectomy) — Appendectomy performed through transumbilical single access laparoscopy, consisting in the removal of the appendix.

SUMMARY:
Laparoscopic appendectomy is a very common intervention in pediatric surgery. To improve outcomes, some teams have developed the use of single-site laparoscopic appendectomy (SILAP). Nevertheless, there is no consensus yet and no published data on the better perioperative analgesia, and different modalities including general intravenous analgesia, locoregional pre-operative analgesia and local analgesia can be used.

DETAILED DESCRIPTION:
The aim of this retrospective study is to describe the different types of perioperative analgesia routinely used and to compare them to determine the more efficient one for early postoperative pain relief.

ELIGIBILITY:
Inclusion Criteria:

* All patients operated on for appendectomy by SILAP, aged 15 years and under in our pediatric surgical center.

Exclusion Criteria:

* Patients aged 16 years or more.
* Patients with concomitant pathologies potentially inducing hyper- or hypoesthesia (e.g. cancers, spinal cord injury, etc...)
* Patients with contraindications for the use of IV analgesics.
* patients operated on for appendectomy through 3-ports laparoscopy or open surgery.
* Opposition of the patients and their representative to the study.

Ages: 1 Day to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All pediatric patients operated on by single-site access for laparoscopic appendectomy.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-08-31 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the level of pain after SILAP during the 24 first hours after surgery. | Up to 16 years of age. From the date of surgery until the end of hospital stay, assessed up to 16 years of age
  Objectified by the quantity of level 2-3 (in morphin equivalent) analgesic used up to 24 hours after surgery.

SECONDARY OUTCOMES:
To assess the level of pain as measured by the different pain scales routinely used. | Up to 16 years of age. From the date of surgery until the end of hospital stay, assessed up to 16 years of age
  Objectified by the higher level of pain quoted during the first 24 hours after surgery.
To assess the level of pain during the initial post-operative recovery room stay. | Up to 16 years of age. From the date of surgery until the end of hospital stay, assessed up to 16 years of age
  Objectified by the higher level of pain quoted during the first 24 hours after surgery and by the amount of level 2-3 analgesic used.
To assess the level of pain after the 24 first hours and until hospital release. | Up to 16 years of age. From the date of surgery until the end of hospital stay, assessed up to 16 years of age
  Objectified by the higher level of pain quoted from 24 hours post-operative to hospital discharge, and by the amount of level 2-3 analgesic used.
To assess the different peri-operative local and loco-regional analgesia modalities used and to compare their efficiency. | Up to 16 years of age. From the date of surgery until the end of hospital stay, assessed up to 16 years of age
  Objectified by the amount of level 2-3 analgesics used in post-operative recovery room and during hospital stay.
To assess the types and gravity of peri-operative and post-analgesia complications. | Up to 16 years of age. From the date of surgery until the end of hospital stay, assessed up to 16 years of age
  Objectified by the description of complications encountered and classified with the Clavien and Dindo gravity scale for surgical complications.

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Schmitt, MD, PhD, Principal Investigator — University hospital of Angers
Locations (1):
- Angers University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goodman LF, Lin AC, Sacks MA, McRae JJLH, Radulescu A, Khan FA. Single site versus conventional laparoscopic appendectomy: some pain for no gain? J Surg Res. 2021 Aug;264:321-326. doi: 10.1016/j.jss.2021.03.010. Epub 2021 Apr 10. PMID 33848830
- [Background] Binet A, Braik K, Lengelle F, Laffon M, Lardy H, Amar S. Laparoscopic one port appendectomy: Evaluation in pediatric surgery. J Pediatr Surg. 2018 Nov;53(11):2322-2325. doi: 10.1016/j.jpedsurg.2017.12.018. Epub 2017 Dec 27. PMID 29370892